CLINICAL TRIAL: NCT03671174
Title: A Three-arm, Multicenter, Open-label Randomized Controlled Trial of Hydroxychloroquine and Low-dose Prednisone on Recurrent Spontaneous Abortion With Undifferentiated Connective Tissue Diseases: Protocol for the Immunosuppressant Regimens for Living FEtuses (ILIFE) Trial
Brief Title: Immunosuppressant Regimens for Living Fetuses Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); China-Japan Union Hospital, Jilin University (Other); Wuxi No. 2 People's Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Liangjing Lu, Professor, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILIFE Study
Record Dates: First submitted 2018-08-30; First posted 2018-09-14 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Undifferentiated Connective Tissue Disease; Recurrent Pregnancy Loss
MeSH Terms: conditions — Undifferentiated Connective Tissue Diseases | interventions — Prednisone; Hydroxychloroquine; Aspirin; Heparin, Low-Molecular-Weight; Enoxaparin; Dalteparin; Nadroparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Prednisone + hydroxychloroquine + anticoagulation (Experimental): Oral low-dose prednisone PLUS Oral hydroxychloroquine PLUS Oral low-dose aspirin PLUS subcutaneous low-molecular-weight heparin
  Interventions: Drug: Prednisone; Drug: Hydroxychloroquine; Drug: Aspirin; Drug: low molecular weight heparin
- Hydroxychloroquine + anticoagulation (Experimental): Oral hydroxychloroquine PLUS Oral low-dose aspirin PLUS subcutaneous low-molecular-weight heparin
  Interventions: Drug: Hydroxychloroquine; Drug: Aspirin; Drug: low molecular weight heparin
- Anticoagulation (Active Comparator): Oral low-dose aspirin PLUS subcutaneous low-molecular-weight heparin
  Interventions: Drug: Aspirin; Drug: low molecular weight heparin

INTERVENTIONS:
Drug: Prednisone — 10mg once daily orally
  Arms: Prednisone + hydroxychloroquine + anticoagulation
Drug: Hydroxychloroquine — 100mg to 200mg twice daily orally
  Arms: Hydroxychloroquine + anticoagulation; Prednisone + hydroxychloroquine + anticoagulation
Drug: Aspirin — 50mg once daily orally
Drug: low molecular weight heparin — Enoxaparin 40mg once daily subcutaneous or dalteparin 5000IU once daily subcutaneous or nadroparin calcium 4100U once daily subcutaneous
  Other Names: Enoxaparin; Dalteparin; Nadroparin

SUMMARY:
Undifferentiated connective tissue diseases (UCTD) are known to increase the risk of pregnancy morbidities, including recurrent pregnancy loss. However, there is no consensus or guideline about the treatment for recurrent pregnancy loss in UCTD patients. Therefore, based on the tendency to thrombosis formation and placental inflammation in the pathogenesis of UCTD, this trial proposes to evaluate the effect of hydroxychloroquine with or without prednisone combined with anticoagulation on pregnancy outcomes in recurrent pregnancy loss patients with UCTD.

DETAILED DESCRIPTION:
Objective: To evaluate the effect of anticoagulation with or without immunomodulatory therapy on pregnancy outcomes of recurrent pregnancy loss with undifferentiated connective tissue diseases Design: a multi-center, randomised, open-label, paralleled study. Patients: Pregnant patients with recurrent pregnancy loss and undifferentiated connective tissue diseases without any known etiology for pregnancy loss (detailed in section 10).

Methods: 420 selected patients are divided into 3 parallel groups (detailed in section 8).

Randomization: Patients who present to relevant clinics for management of recurrent spontaneous abortion (RSA) will be evaluated for inclusion criteria and exclusion criteria by a formed physician. Once patient is eligible for the study, the co-investigator will obtain written patient's consent. Participants will be randomized into one of the 3 groups. Randomized numbers will be generated by pharmacology research personnel in Renji Hospital. Given the different administrated medications, neither the patient nor the provider will be blinded.

Follow-up: Consultation will be scheduled every 4 weeks from confirmed pregnancy until delivery. The co-investigator will complete a follow-up survey including clinical, biological data.

Missing data: Patients are willing to drop the study, unavailable, incompliant, with severe complications or with severe adverse effects. The missing data will be recorded in detail and be analysed with last pregnancy outcome.

ELIGIBILITY:
Inclusion criteria

Women who meet the following inclusion criteria will be eligible to participate in the study:

1. At reproductive age (20-40 years old).
2. Trying to conceive.
3. Diagnosed with UCTD[2]: at least one symptoms or signs suggesting connective tissue disease(CTD) and with at least one presence of auto-antibodies, including antinuclear antibody (ANA), anti-SSA antibody, while not fulfilling any classification criteria of a defined CTD.
4. Diagnosed with RSA[39]: two or more failed pregnancies of unknown origin.
5. Providing written informed consent. Exclusion criteria

Women who meet any of the following criteria will be excluded from the study:

1.Any known etiology of previous pregnancy loss:

1. Diagnosis of antiphospholipid antibody syndrome.
2. Known paternal, maternal or embryo chromosome abnormality.
3. Maternal endocrine dysfunction: corpus luteal insufficiency; polycystic ovarian syndrome; premature ovarian failure (follicle stimulating hormone, FSH ≥20uU/L in follicular phase); hyperprolactinemia; thyroid disease; diabetes mellitus; other hypothalamic-pituitary-adrenal axis abnormality.
4. Maternal anatomical abnormality: uterine malformation; Asherman syndrome; cervical incompetence; uterine fibrosis more than 5 cm.
5. Vaginal infection. 2.Any known severe cardiac, hepatic, renal, hematological or endocrinal diseases:

(1)Alanine transaminase (ALT) or aspartate transaminase(AST) more than twice the upper limit of normal.

(2)Clearance of creatinine less than 30mL/min. (3)Leucocytes less than 2.5*10^9/L, or Hemoglobine less than 85g/L, or Platelet less than 50~10^9/L.

3.Any active infection:

1. Active viral hepatitis including hepatitis B virus (HBV), hepatitis C virus (HCV).
2. Active infection including V aricella-zostervirus(VZV), human immunodeficiency virus (HIV), syphilis or tuberculosis.

4.Allergic to prednisone, hydroxychloroquine, low-molecular-weight heparin or aspirin.

5.Disease history as follows:

1. Past history of digestive ulcers or upper gastrointestinal hemorrhage.
2. Past history of malignancy.
3. Past history of epilepsia or psychotic disorders. 6.Woman unable to consent or impossible to follow-up.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 420 (Estimated)
Dates: Start 2019-08-02 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | After 28 weeks of gestation
  Percentage of all cycles that lead to live birth

SECONDARY OUTCOMES:
Rate of miscarriage | Within 28 weeks of gestation
  Spontaneous pregnancy loss within 28 weeks of gestation, confirmed by pelvic ultrasound findings. This includes no yolk sac or embryo in a gestational sac and an embryo without cardiac activity.
Premature birth | between 28 and 37 weeks of gestations
  live birth between 28 and 37 weeks of gestations Prematurity (live birth between 28 and 37 weeks of gestations); Eclampsia (new-onset hypertension after 20 weeks of gestation, +/- proteinuria > 300mg/24h, with or without any organ damage with seizures); Fetal abnormality (congenital heart conduction block, neonatal lupus or malformation)
Intrauterine growth retardation | between 28 and 37 weeks of gestations
  weight below the 10th percentile for the gestational age Prematurity (live birth between 28 and 37 weeks of gestations); Eclampsia (new-onset hypertension after 20 weeks of gestation, +/- proteinuria > 300mg/24h, with or without any organ damage with seizures); Fetal abnormality (congenital heart conduction block, neonatal lupus or malformation)
Gestational age and weight at birth | post-partum 6 weeks
  the children's gestational age and weight at birth
Survival at 28 days | post-partum 6 weeks
  still alive at 28 days
Number of newborns with treatment-related adverse events assessed by 3 parameters | post-partum 6 weeks
  assess the number of the newborns with abnormal vision, hearing and length at 6 weeks
Congenital abnormality | post-partum 6 weeks
  congenital heart conduction block, neonatal lupus or malformation
Eclampsia | After 20 weeks of gestation
  New-onset hypertension after 20 weeks of gestation, with or without proteinuria > 300mg/24h, with or without any organ damage with seizures
Number of participants with Infection | through study completion, an average of 1.5 years
  Infection of respiratory tract, digestive tract, urinary tract and skin
Gestational diabetes mellitus | through study completion, an average of 1.5 years
  Clinical diagnosis of gestational diabetes mellitus
Activity of UCTD | through study completion, an average of 1.5 years
  New onset or aggravation of symptoms like arthritis, rash, Reynolds phenomenon, proteinuria, etc.
Number of participants who evolved to systemic lupus erythematosus(SLE) from undifferentiated connective tissue diseases(UCTD) | post-partum 6 weeks
  Clinical diagnosis of systemic lupus erythematosus
Number of participants who evolved to Sjogren's syndrome(SS) from undifferentiated connective tissue diseases(UCTD) | post-partum 6 weeks
  Clinical diagnosis of Sjogren's syndrome
Number of participants who evolved to systemic sclerosis(SSc) from undifferentiated connective tissue diseases(UCTD) | post-partum 6 weeks
  Clinical diagnosis of systemic sclerosis
Number of participants who evolved to polymyositis(PM) or dermatomyositis(DM) from undifferentiated connective tissue diseases(UCTD) | post-partum 6 weeks
  Clinical diagnosis of polymyositis or dermatomyositis
Number of participants who evolved to antiphospholipid syndrome (APS) from undifferentiated connective tissue diseases(UCTD) | post-partum 6 weeks
  Clinical diagnosis of antiphospholipid syndrome
Number of participants who evolved to rheumatoid arthritis (RA) from undifferentiated connective tissue diseases(UCTD) | post-partum 6 weeks
  Clinical diagnosis of rheumatoid arthritis
Number of participants who evolved to mixed connective tissue disease(MCTD) from undifferentiated connective tissue diseases(UCTD) | post-partum 6 weeks
  Clinical diagnosis of mixed connective tissue disease

CONTACTS AND LOCATIONS:
Overall Officials: Liangjing Lu, Study Chair — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mosca M, Neri R, Bombardieri S. Undifferentiated connective tissue diseases (UCTD): a review of the literature and a proposal for preliminary classification criteria. Clin Exp Rheumatol. 1999 Sep-Oct;17(5):615-20. PMID 10544849
- [Background] Andreoli L, Bertsias GK, Agmon-Levin N, Brown S, Cervera R, Costedoat-Chalumeau N, Doria A, Fischer-Betz R, Forger F, Moraes-Fontes MF, Khamashta M, King J, Lojacono A, Marchiori F, Meroni PL, Mosca M, Motta M, Ostensen M, Pamfil C, Raio L, Schneider M, Svenungsson E, Tektonidou M, Yavuz S, Boumpas D, Tincani A. EULAR recommendations for women's health and the management of family planning, assisted reproduction, pregnancy and menopause in patients with systemic lupus erythematosus and/or antiphospholipid syndrome. Ann Rheum Dis. 2017 Mar;76(3):476-485. doi: 10.1136/annrheumdis-2016-209770. Epub 2016 Jul 25. PMID 27457513
- [Background] Spinillo A, Beneventi F, Caporali R, Ramoni V, Montecucco C. Undifferentiated connective tissue diseases and adverse pregnancy outcomes. An undervalued association? Am J Reprod Immunol. 2017 Dec;78(6). doi: 10.1111/aji.12762. Epub 2017 Sep 16. PMID 28921728
- [Result] Alarcon GS, Williams GV, Singer JZ, Steen VD, Clegg DO, Paulus HE, Billingsley LM, Luggen ME, Polisson RP, Willkens RF, et al. Early undifferentiated connective tissue disease. I. Early clinical manifestation in a large cohort of patients with undifferentiated connective tissue diseases compared with cohorts of well established connective tissue disease. J Rheumatol. 1991 Sep;18(9):1332-9. PMID 1757934
- [Result] Laczik R, Soltesz P, Szodoray P, Szekanecz Z, Kerekes G, Paragh G, Rajnavolgyi E, Abel G, Szegedi G, Bodolay E. Impaired endothelial function in patients with undifferentiated connective tissue disease: a follow-up study. Rheumatology (Oxford). 2014 Nov;53(11):2035-43. doi: 10.1093/rheumatology/keu236. Epub 2014 Jun 10. PMID 24917564
- [Result] Spinillo A, Beneventi F, Locatelli E, Ramoni V, Caporali R, Alpini C, Albonico G, Cavagnoli C, Montecucco C. The impact of unrecognized autoimmune rheumatic diseases on the incidence of preeclampsia and fetal growth restriction: a longitudinal cohort study. BMC Pregnancy Childbirth. 2016 Oct 18;16(1):313. doi: 10.1186/s12884-016-1076-8. PMID 27756248
- [Result] Mosca M, Neri R, Strigini F, Carmignani A, Totti D, Tavoni A, Bombardieri S. Pregnancy outcome in patients with undifferentiated connective tissue disease: a preliminary study on 25 pregnancies. Lupus. 2002;11(5):304-7. doi: 10.1191/0961203302lu187oa. PMID 12090565
- [Result] Spinillo A, Beneventi F, Epis OM, Montanari L, Mammoliti D, Ramoni V, Di Silverio E, Alpini C, Caporali R, Montecucco C. The effect of newly diagnosed undifferentiated connective tissue disease on pregnancy outcome. Am J Obstet Gynecol. 2008 Dec;199(6):632.e1-6. doi: 10.1016/j.ajog.2008.05.008. Epub 2008 Jul 29. PMID 18667193
- [Result] Alijotas-Reig J, Ferrer-Oliveras R; EUROAPS Study Group. The European Registry on Obstetric Antiphospholipid Syndrome (EUROAPS): a preliminary first year report. Lupus. 2012 Jun;21(7):766-8. doi: 10.1177/0961203312440058. PMID 22635227
- [Result] Proietta M, Ferrero S, Ferri L, Cifani N, Bruno G, Del Porto F. Recurrent miscarriages in women not fulfilling classification criteria for antiphospholipid antibody syndrome. Int J Immunopathol Pharmacol. 2014 Jul-Sep;27(3):429-32. doi: 10.1177/039463201402700313. PMID 25280034
- [Result] Vaz CC, Couto M, Medeiros D, Miranda L, Costa J, Nero P, Barros R, Santos MJ, Sousa E, Barcelos A, Ines L. Undifferentiated connective tissue disease: a seven-center cross-sectional study of 184 patients. Clin Rheumatol. 2009 Aug;28(8):915-21. doi: 10.1007/s10067-009-1175-2. Epub 2009 Apr 24. PMID 19390908
- [Result] Bansal AS. Joining the immunological dots in recurrent miscarriage. Am J Reprod Immunol. 2010 Nov;64(5):307-15. doi: 10.1111/j.1600-0897.2010.00864.x. PMID 20528832
- [Result] Tempfer CB, Kurz C, Bentz EK, Unfried G, Walch K, Czizek U, Huber JC. A combination treatment of prednisone, aspirin, folate, and progesterone in women with idiopathic recurrent miscarriage: a matched-pair study. Fertil Steril. 2006 Jul;86(1):145-8. doi: 10.1016/j.fertnstert.2005.12.035. Epub 2006 May 23. PMID 16716321
- [Result] Gomaa MF, Elkholy AG, El-Said MM, Abdel-Salam NE. Combined oral prednisolone and heparin versus heparin: the effect on peripheral NK cells and clinical outcome in patients with unexplained recurrent miscarriage. A double-blind placebo randomized controlled trial. Arch Gynecol Obstet. 2014 Oct;290(4):757-62. doi: 10.1007/s00404-014-3262-0. Epub 2014 May 13. PMID 24818590
- [Result] Gonzalez-Lopez L, Gamez-Nava JI, Jhangri G, Russell AS, Suarez-Almazor ME. Decreased progression to rheumatoid arthritis or other connective tissue diseases in patients with palindromic rheumatism treated with antimalarials. J Rheumatol. 2000 Jan;27(1):41-6. PMID 10648016
- [Result] Clowse ME, Magder L, Witter F, Petri M. Hydroxychloroquine in lupus pregnancy. Arthritis Rheum. 2006 Nov;54(11):3640-7. doi: 10.1002/art.22159. PMID 17075810
- [Result] Koh JH, Ko HS, Kwok SK, Ju JH, Park SH. Hydroxychloroquine and pregnancy on lupus flares in Korean patients with systemic lupus erythematosus. Lupus. 2015 Feb;24(2):210-7. doi: 10.1177/0961203314555352. Epub 2014 Oct 10. PMID 25305214
- [Result] Luo Y, Zhang L, Fei Y, Li Y, Hao D, Liu Y, Zhao Y. Pregnancy outcome of 126 anti-SSA/Ro-positive patients during the past 24 years--a retrospective cohort study. Clin Rheumatol. 2015 Oct;34(10):1721-8. doi: 10.1007/s10067-015-3050-7. Epub 2015 Aug 26. PMID 26384980
- [Result] Sciascia S, Hunt BJ, Talavera-Garcia E, Lliso G, Khamashta MA, Cuadrado MJ. The impact of hydroxychloroquine treatment on pregnancy outcome in women with antiphospholipid antibodies. Am J Obstet Gynecol. 2016 Feb;214(2):273.e1-273.e8. doi: 10.1016/j.ajog.2015.09.078. Epub 2015 Sep 30. PMID 26429521
- [Result] Izmirly PM, Kim MY, Llanos C, Le PU, Guerra MM, Askanase AD, Salmon JE, Buyon JP. Evaluation of the risk of anti-SSA/Ro-SSB/La antibody-associated cardiac manifestations of neonatal lupus in fetuses of mothers with systemic lupus erythematosus exposed to hydroxychloroquine. Ann Rheum Dis. 2010 Oct;69(10):1827-30. doi: 10.1136/ard.2009.119263. Epub 2010 May 6. PMID 20447951
- [Derived] Yang S, Ni R, Lu Y, Wang S, Xie F, Zhang C, Lu L. A three-arm, multicenter, open-label randomized controlled trial of hydroxychloroquine and low-dose prednisone to treat recurrent pregnancy loss in women with undifferentiated connective tissue diseases: protocol for the Immunosuppressant regimens for LIving FEtuses (ILIFE) trial. Trials. 2020 Sep 9;21(1):771. doi: 10.1186/s13063-020-04716-1. PMID 32907619